CLINICAL TRIAL: NCT00234156
Title: Sensitivity to Fructose-Induced Palmitate Synthesis in End-Stage Renal Disease
Brief Title: The Effect of Fructose on Blood Fats in Dialysis Patients and Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Robert C. Atkins Foundation (Other); The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RUH IRB #LHU 0471
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: End-stage Renal Disease
Keywords: Fructose; Lipogenesis; Triglycerides; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Fructose; Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- renal disease (Active Comparator): High fat diet: The composition will be: 35% of energy as fat, 50% carbohydrate, 15% protein (~1.3 g/kg), sat:mono:poly 1:3:1, cholesterol 200 mg/d, 30% starch,15% sugar, 3% fructose, and 25 gm fiber/d. This relatively high fat diet, which falls within the recommendations by the National Kidney Foundation for hemodialysis patients, will suppress fatty acid synthesis in normal volunteers.
  Fructose in 360 ml water will be orally administered as 1.4 g/kg (~100 g or 400 kcal for a 70 kg person), divided into 30 mL (1 ounce) doses given every 1/2h for 6 hours.
  Interventions: Procedure: oral fructose and high fat diet
- normal (Active Comparator): High fat diet: The composition will be: 35% of energy as fat, 50% carbohydrate, 15% protein (~1.3 g/kg), sat:mono:poly 1:3:1, cholesterol 200 mg/d, 30% starch,15% sugar, 3% fructose, and 25 gm fiber/d. This relatively high fat diet, which falls within the recommendations by the National Kidney Foundation for hemodialysis patients, will suppress fatty acid synthesis in normal volunteers.
  Fructose in 360 ml water will be orally administered as 1.4 g/kg (~100 g or 400 kcal for a 70 kg person), divided into 30 mL (1 ounce) doses given every 1/2h for 6 hours.
  Interventions: Procedure: oral fructose and high fat diet

INTERVENTIONS:
Procedure: oral fructose and high fat diet — High fat diet: The composition will be: 35% of energy as fat, 50% carbohydrate, 15% protein (~1.3 g/kg), sat:mono:poly 1:3:1, cholesterol 200 mg/d, 30% starch,15% sugar, 3% fructose, and 25 gm fiber/d. This relatively high fat diet, which falls within the recommendations by the National Kidney Foundation for hemodialysis patients, will suppress fatty acid synthesis in normal volunteers.
  Fructose in 360 ml water will be orally administered as 1.4 g/kg (~100 g or 400 kcal for a 70 kg person), divided into 30 mL (1 ounce) doses given every 1/2h for 6 hours.

SUMMARY:
This study will evaluate how a common dietary sugar (fructose) raises blood fats (triglycerides). We will determine whether the production of fat from fructose is higher in dialysis patients compared to healthy volunteers. Dialysis patients have high levels of hormone-like substances called cytokines that may increase blood fats. The results will help set better guidelines for diets for the general population and patients with kidney disease who are at high risk for heart attack and stroke.

There will be one or two outpatient screening visit(s) and a one-week (6 nights) stay at the Rockefeller University Hospital.

DETAILED DESCRIPTION:
Fifteen hemodialysis patients and 15 healthy volunteers will be studied.

Outpatient screening visit(s): consent, fasting blood and urine analysis, a physical exam, an EKG and a 2-hour oral glucose tolerance test to screen for diabetes.

Inpatient admission:

* Standardized diet that follows the guidelines for hemodialysis patients and healthy volunteers to maintain a stable weight.
* Blood and urine sampling. The total amount of blood drawn is less than 1 cup.
* To measure the production of fat from fructose, a trace amount of a non-radioactive labeled precursor of fat (13C-acetate) will be infused through a venous catheter for 22 hours.

At the end of the infusion, a sweet drink (fructose in 1 ounce of water) will be given orally every half hour for 6 hours.

• Two small samples of fat taken right below the skin will be obtained after injection of a small amount of numbing medicine into the abdominal and gluteal regions.

Dialysis patients will receive their usual dialysis at The Rogosin Institute Manhattan, Brooklyn or Queens Dialysis Units.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, 18-75 years of age.
2. Chronic renal failure with hemodialysis 3x/week for at least 6 months and adequate dialysis as judged by a nephrologist who is not a study investigator.
3. Fasting TG <600 mg/dl, LDL cholesterol <190 mg/dl (off lipid-lowering medication)
4. Willing and able to change Renagel, a noncalcemic phosphate binder (poly[allylamine hydrochloride]) which has LDL-lowering effects, to the same amount of another phosphate binder for 1 month prior to the screening visit until the completion of the study.
5. Willing and able to temporarily stop Sensipar (cinacalcet) for 1 week before the study admission until completion of the study (a total of ~2 weeks).
6. Willing and able to stop ASA (except low dose ASA in patients with vascular disease), NSAID, fish oil, psyllium, other nonprescribed vitamins/supplements for 1 week prior to study until completion of study.
7. Willing and able to sign an informed consent.
8. Willing to refrain from participation in an investigational drug study for the duration of the study.

Exclusion Criteria:

1. Diabetes (fasting blood sugar >126 twice or an abnormal 2 hour OGTT)
2. Unstable clinical condition, including acute febrile illness within 1 month of admission
3. Chronic infection, including hepatitis and HIV infection
4. Gastrointestinal disease resulting in significant GI dysfunction or malabsorption
5. Lipid-lowering medication
6. Mean systolic blood pressure >180 or diastolic pressure >110 taken immediately before 6 dialysis treatments over the 2 weeks before the screening visit 7/15/2008 Form version 6/13/2005 #LHU-0471-0407 Page 8of 16f
7. BMI >35 (markedly obese)
8. Hemoglobin <10.0
9. Prednisone, estrogen/progesterone, other steroids, Synthroid, endocrine disease
10. Coumadin and an INR >1.5
11. Cigarette smoking >1/2 pack/day
12. Abuse of ethanol (greater than 2 drinks/day) or illicit drugs
13. If female, pregnant or breast feeding
14. Participation in a study of an investigational drug during the 30 days preceding the start of the screening period
15. Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study

Healthy Controls:

Inclusion Criteria

1. Male and females, 18-75 years of age 2. LDL <160 mg/dl, HDL-C >30 mg/dl, TG <250 mg/dl 3. Willing and able to stop ASA, NSAID, fish oil, psyllium, other vitamins/supplements for 1 week prior to study until completion of study 4. Willing and able to sign an informed consent 5. Willing to refrain from participation in an investigational drug study for the duration of the study Exclusion Criteria

1. Systemic illnesses, including diabetes (FBS >126 twice or abnormal OGTT), cardiovascular disease, hepatitis, endocrine disease, HIV infection.
2. Prescription medications, including contraceptives.
3. Acute febrile illness within 1 month of admission.
4. BMI >35 (markedly obese) or>10% below maximum weight.
5. Weight change of >10% usual weight in the previous 6 months.
6. Blood pressure >140/90.
7. HB <11 female, <12 male.
8. CRP >5.0 on 2 occasions. 7/15/2008 Form version 6/13/2005 #LHU-0471-0407 Page 9of 16f
9. Abuse of ethanol (greater than 2 drinks/day) or illicit drugs.
10. Cigarette smoking >1/2 pack/day.
11. Unusual diet or extreme physical activity (e.g. marathon runner).
12. If female, pregnant or breast feeding.
13. Participation in a study of an investigational drug during the 30 days preceding the start of the screening period.
14. Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Peak percent de novo palmitate in blood triglycerides after oral fructose | day 1 and day 6

SECONDARY OUTCOMES:
Relationship between TNF and/or its soluble receptors and % newly formed palmitate | Day 1 and Day 6
fatty acid composition of TG and adipose tissue | Day 1 of hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C. Hudgins, MD, Principal Investigator — Rockefeller University, Rogosin Institute
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Hudgins LC, Parker TS, Levine DM, Hellerstein MK. A dual sugar challenge test for lipogenic sensitivity to dietary fructose. J Clin Endocrinol Metab. 2011 Mar;96(3):861-8. doi: 10.1210/jc.2010-2007. Epub 2011 Jan 20. PMID 21252253